CLINICAL TRIAL: NCT05822635
Title: Intraoperative Endoscopy Using a Thin, Single-Use, Flexible Cholangiopancreatoscope
Brief Title: SpyGlass Surgical Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7161
Record Dates: First submitted 2023-04-07; First posted 2023-04-21 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Diseases; Bile Duct Diseases; Hepatic Disease
MeSH Terms: conditions — Pancreatic Diseases; Bile Duct Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects with complex pancreaticobiliary disease: All subjects will undergo the intraoperative endoscopy with either the SpyGlass Discover System or the SpyGlass DS Direct Visualization System.
  Interventions: Device: SpyGlass Discover Digital System or SpyGlass DS Direct Visualization System

INTERVENTIONS:
Device: SpyGlass Discover Digital System or SpyGlass DS Direct Visualization System — Observational, prospective study for the clinical utility of the SpyGlass Discover Digital Catheter and the SpyScope DS Catheter during an intraoperative endoscopy procedure.

SUMMARY:
* To document the clinical utility of diagnostic and/or therapeutic intraoperative endoscopy using a thin, single-use, flexible cholangiopancreatoscope
* To identify specific surgical procedures in which intraoperative use of a thin, single use, flexible cholangiopancreatoscope suggests clinically meaningful benefit and generate a hypothesis for possible subsequent claims-supportive study

DETAILED DESCRIPTION:
This case series aims to document the clinical utility of intraoperative endoscopy using a thin, disposable, flexible cholangiopancreatoscope in procedures including but not limited to:

* Evaluation of biliary lesion(s) during surgical management of common bile duct (CBD) and intrahepatic duct (IHD) strictures, with or without biopsy
* Transcystic/transcholedochal clearance of biliary stone(s)/sludge/cast with or without mechanical, electrohydraulic or laser lithotripsy
* Treatment of hepatolithiasis
* Assessment of communication between the biliary tree and the cyst in the setting of ruptured hydatid parasitic cysts or abcesses
* Visualization of intraductal papillary mucinous neoplasm (IPMN) lesion(s) with or without biopsy
* Assessment of pancreatic duct (PD) strictures in chronic pancreatitis, with or without biopsy

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for intraoperative endoscopy using a thin, single-use, flexible cholangiopancreatoscope
* Written informed consent from patient or legally authorized representative of the patient

Exclusion Criteria:

* Contraindication for intraoperative endoscopy using a thin, single-use, flexible cholangiopancreatoscope
* <18 years of age
* Potentially vulnerable subjects, including, but not limited to pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complex pancreaticobiliary disease
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Technical success | During study procedure
  Perform intraoperative endoscopy as intended using a thin, single-use, flexible cholangiopancreatoscope as desired, including but not limited to:
  * Direct visualization of target lesion or stricture
  * Obtaining biopsies
  * Initiating and/or completing stone clearance

SECONDARY OUTCOMES:
Number of adverse events | 1 month
  Serious adverse events related to the study device, accessory devices used throughout the working channel of the SpyGlass™ system, or the intraoperative endoscopy procedure
Endoscopist rating of clinical impact of study procedure | During study procedure
  Characterization and rating of the clinical benefit and impact of intraoperative endoscopy using a thin, single-use, flexible cholangiopancreatoscope to the surgical procedure on a 1 (highly dissatisfied) to 10 (highly satisfied) scale
Adequate diagnostic yield | 1 month
  Adequate diagnostic yield of tissue biopsy for histopathology assessment
Endoscopist rating of device | During study procedure
  Rating of the intraoperative performance of the SpyGlass™ system and accessories during intraoperative endoscopy procedure compared to marketed reusable endoscopes on a 1 (highly dissatisfied) to 10 (highly satisfied) scale:
  1. Image quality
  2. Ability to irrigate field of view through the irrigation channels
  3. Ability to aspirate through the working channel
  4. Ability to retroflex
  5. Ability to obtain targeted biopsies using biopsy forceps
  6. Ability to grasp stones using wire basket
  7. Ability to perform lithotripsy
  8. Ability to advance accessories through catheter
  9. Ability to selectively advance into targeted ducts

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Indiana University Health, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
- Lanzhou University No. 1 Hospital, Lanzhou, Gansu, China
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No